CLINICAL TRIAL: NCT06544668
Title: A Clinical Study to Establish a Dynamic Prediction Model for Bone Metastases Based on Breast Cancer Real-world Data
Brief Title: A Study for Dynamic Prediction Model of Breast Cancer Bone Metastases
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC4673
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Bone Metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients with bone metastasis
  Interventions: Other: Breast cancer patients with bone metastasis
- Breast cancer patients without bone metastasis
  Interventions: Other: Breast cancer patients without bone metastasis

INTERVENTIONS:
Other: Breast cancer patients with bone metastasis — This study is an observational study
  Groups: Breast cancer patients with bone metastasis
Other: Breast cancer patients without bone metastasis — This study is an observational study
  Groups: Breast cancer patients without bone metastasis

SUMMARY:
The purpose of this study is to identify the risk factors of bone metastasis in breast cancer patients so as to develop a dynamic prediction model using real world clinical data. The multicenter data will be retrospectively collected, and the clinical characteristics related to bone metastasis will be analyzed.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women worldwide and bones are the most common sites of metastases in breast cancer patients(~70%). Bone metastasis often leads to skeletal-related events (SREs) ,which may not only reduce the quality of life in patients, but also affect the long-term survival. Therefore, early detection and early intervention of bone metastasis are particularly important for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with breast cancer by histopathology;
2. Age between 20 and 70 years old;
3. The first diagnosis time is between 2010 and 2020;
4. Complete diagnosis and treatment information, including basic information, breast cancer diagnosis, surgery, recurrence diagnosis data (including the diagnosis of the metastasis sites), anti-tumor treatment data, bone health and bone metastasis-related diagnosis and treatment data, etc.;
5. Sufficient available follow-up information.

Exclusion Criteria:

1. Missing important basic information (including initial and recurrent pathology, stage, pathological grade and time, surgery time, and drug treatment);
2. With distant metastasis at the initial diagnosis;
3. Patients with autoimmune diseases or aggressive viral infections (such as HIV or hepatitis);
4. Other malignant tumors;
5. Unclear information about distant metastasis.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3500 breast cancer patients diagnosed between 2010 and 2020.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2024-08-06 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
To identify the risk factors and develop a prediction model for bone metastasis in breast cancer patients | 60 months
  The correlation between clinical characteristics and bone metastasis, and the accuracy of prediction model

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No